CLINICAL TRIAL: NCT00769886
Title: A Multi-Center, Double-Masked, Randomized, Vehicle and Active Controlled Evaluation of the Onset and Duration of Action of KetoNaph Ophthalmic Solution in the Conjunctival Allergen Challenge Model of Acute Allergic Conjunctivitis
Brief Title: Ketotifen/Naphazoline Ophthalmic Solution in the Conjunctival Allergen Challenge Model of Allergic Conjunctivitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 571
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2020-10

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Ketotifen; Naphazoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- KetoNaph (Experimental): KetoNaph (ketotifen fumarate 0.025%, naphazoline HCl 0.05%) ophthalmic solution
  Interventions: Drug: Ketotifen/naphazoline
- Naphazoline (Active Comparator): Naphazoline HCl 0.05% ophthalmic solution
  Interventions: Drug: Naphazoline
- Ketotifen (Active Comparator): Ketotifen fumarate 0.025% ophthalmic solution
  Interventions: Drug: Ketotifen
- Vehicle (Placebo Comparator): Vehicle of KetoNaph ophthalmic solution
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Ketotifen/naphazoline — One drop of ketotifen/naphazoline in study eye at visit 3 and visit 4.
  Arms: KetoNaph
Drug: Ketotifen — One drop of Ketotifen in study eye at visit 3 and visit 4.
  Arms: Ketotifen
Drug: Naphazoline — One drop of naphazoline in study eye at vist 3 and visit 4.
  Arms: Naphazoline
Drug: Vehicle — One drop of vehicle in study eye at visit 3 and visit 4.
  Arms: Vehicle

SUMMARY:
The purpose of this study is to establish the safety and efficacy of ketotifen/naphazoline ophthalmic solution compared to vehicle and its individual components in alleviating the signs and symptoms of conjunctival allergen challenge (CAC)-induced allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of ocular allergies and positive skin test reaction to cat hair, cat dander, grasses, ragweed, and/or trees within the past 24 months.
* Calculated best-corrected visual acuity of 0.7 logMAR or better in each eye as measured using the ETDRS chart.
* Positive bilateral conjunctival allergen challenge(CAC)reaction within 10 minutes of instillation of the last titration of allergen at visit 1.
* Positive bilateral CAC reaction in at least 2 out of 3 time points at visit 2.

Exclusion Criteria:

* Known contraindications or sensitivities to the study medication or its components.
* Any ocular condition that, in the opinion of the investigator, could affect the subjects safety or trial parameters.
* Use of disallowed medications during the period indicated prior to study enrollment or during the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Consultants, Inc., North Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Started | 36; 72 Eyes | 36; 72 Eyes | 35; 70 Eyes | 37; 74 Eyes
Completed | 31; 62 Eyes | 32; 64 Eyes | 34; 68 Eyes | 35; 70 Eyes
Not Completed | 5; 10 Eyes | 4; 8 Eyes | 1; 2 Eyes | 2; 4 Eyes

BASELINE CHARACTERISTICS:
Groups:
- KetoNaph: KetoNaph (ketotifen fumarate 0.025%, naphazoline HCl 0.05%) ophthalmic solution Ketotifen/naphazoline: One drop of ketotifen/naphazoline in study eye at visit 3 and visit 4.
- Ketotifen: Ketotifen fumarate 0.025% ophthalmic solution Ketotifen: One drop of Ketotifen in study eye at visit 3 and visit 4.
- Naphazoline: Naphazoline HCl 0.05% ophthalmic solution Naphazoline: One drop of naphazoline in study eye at vist 3 and visit 4.
- Vehicle: Vehicle of KetoNaph ophthalmic solution Vehicle: One drop of vehicle in study eye at visit 3 and visit 4.
- Total: Total of all reporting groups
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle | Total
Number analyzed (Participants) | 36 | 36 | 35 | 37 | 144
Age, Continuous [Mean (Full Range); unit: years] | 33.63 [8 to 63] | 34.15 [10 to 71] | 35.56 [8 to 63] | 33.09 [9 to 71] | 34.10 [8 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 18 | 21 | 77
  Male | 16 | 18 | 17 | 16 | 67

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Ocular itching was evaluated by the participant at 3, 5, and 7 minutes post challenge. Assessments were made using a 0-4 numerical analog scale, allowing 0.5-unit increments (but disallowing 0.25-unit increments), where: 0.0 = None and 4.0 = Incapacitating itch with an irresistible urge to rub.
Time Frame: 3, 5, and 7 minutes post challenge at 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 36 | 36 | 35 | 37
Number analyzed (eyes) | 72 | 71 | 70 | 74
score on a scale
  3 minutes post-challenge | 0.50 (0.835) | 0.49 (0.860) | 1.87 (0.932) | 1.93 (0.998)
  5 minutes post-challenge | 0.56 (0.785) | 0.69 (0.923) | 1.90 (0.936) | 2.17 (0.885)
  7 minutes post-challenge | 0.56 (0.856) | 0.72 (0.885) | 1.75 (0.971) | 1.97 (0.984)

2. Primary Outcome: Conjunctival Hyperemia
Description: Conjunctival hyperemia was evaluated by the Investigator at 7, 15, and 20 minutes post challenge. Assessments were completed using a 0-4 numerical analog scale, allowing 0.5-unit increments, where: 0.0 = None and 4.0 = Extremely severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 36 | 36 | 35 | 37
Number analyzed (eyes) | 72 | 71 | 70 | 74
units on a scale
  7 minutes post-challenge | 1.13 (0.872) | 1.49 (0.761) | 1.62 (0.860) | 2.24 (0.581)
  15 minutes post-challenge | 1.39 (0.865) | 1.89 (0.712) | 1.68 (0.957) | 2.33 (0.551)
  20 minutes post-challenge | 1.26 (0.818) | 1.77 (0.805) | 1.53 (0.959) | 2.24 (0.587)

3. Secondary Outcome: Ciliary Redness
Description: Ciliary hyperemia (redness) was evaluated by the Investigator at 7, 15, and 20 minutes post challenge. Assessments were made using a 0-4 scale, allowing 0.5- unit increments, with 0.0 = None and 4.0 = Extremely severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: This outcome measure was not assessed for the Vehicle group.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 36 | 36 | 35 | 0
Number analyzed (eyes) | 72 | 71 | 70 | 0
units on a scale
  7 minutes post-challenge | 1.05 (0.873) | 1.39 (0.774) | 1.66 (0.917) |
  15 minutes post-challenge | 1.28 (0.907) | 1.79 (0.791) | 1.71 (0.995) |
  20 minutes post-challenge | 1.15 (0.854) | 1.77 (0.810) | 1.58 (1.032) |

4. Secondary Outcome: Episcleral Redness
Description: Episcleral hyperemia (redness) was evaluated by the Investigator at 7, 15, and 20 minutes post challenge. Assessments were made using a 0-4 scale, allowing 0.5- unit increments, with 0.0 = None and 4.0 = Extremely severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: This outcome measure was not assessed for the Vehicle group.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 36 | 36 | 35 | 0
Number analyzed (eyes) | 72 | 71 | 70 | 0
score on a scale
  7 minutes post-challenge | 1.21 (0.891) | 1.52 (0.749) | 1.71 (0.951) |
  15 minutes post-challenge | 1.41 (0.865) | 1.87 (0.732) | 1.77 (0.988) |
  20 minutes post-challenge | 1.35 (0.895) | 1.88 (0.777) | 1.68 (1.026) |

5. Secondary Outcome: Chemosis
Description: Chemosis was evaluated by the Investigator at 7, 15, and 20 minutes post challenge on a 0-4 numerical analog scale, allowing 0.5-unit increments, where: 0.0 = None and 4.0 = Extremely severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: This outcome measure was not assessed for the Vehicle group.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 36 | 36 | 35 | 0
Number analyzed (eyes) | 72 | 71 | 70 | 0
score on a scale
  7 minutes post-challenge | 0.22 (0.410) | 0.22 (0.313) | 0.51 (0.705) |
  15 minutes post-challenge | 0.29 (0.488) | 0.42 (0.420) | 0.66 (0.787) |
  20 minutes post-challenge | 0.34 (0.549) | 0.41 (0.450) | 0.66 (0.869) |

6. Secondary Outcome: Eyelid Swelling
Description: Lid swelling was evaluated by the subject at 7, 15, and 20 minutes post challenge on a 0- 3 numerical analog scale, with 0.5-unit increments disallowed, where: 0.0 = None and 3.0 = Severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: This outcome measure was not assessed for the Vehicle group.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 36 | 36 | 35 | 0
Number analyzed (eyes) | 72 | 71 | 70 | 0
score on a scale
  7 minutes post-challenge | 0.13 (0.373) | 0.32 (0.604) | 0.61 (0.783) |
  15 minutes post-challenge | 0.25 (0.550) | 0.37 (0.638) | 0.61 (0.746) |
  20 minutes post-challenge | 0.26 (0.581) | 0.39 (0.686) | 0.59 (0.729) |

7. Secondary Outcome: Percentage of Eyes With Tearing
Description: Tearing was evaluated by the subject at 7, 15, and 20 minutes post challenge (absent or present). Tearing was recorded as either absent or present.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: This outcome measure was not assessed for the Vehicle group.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 36 | 36 | 35 | 0
Number analyzed (eyes) | 72 | 71 | 70 | 0
eyes
  7 minutes post-challenge | 3 | 11 | 23 |
  15 minutes post-challenge | 6 | 7 | 16 |
  20 minutes post-challenge | 5 | 7 | 13 |

8. Secondary Outcome: Percentage of Eyes With Ocular Mucus Drainage
Description: Ocular mucous discharge was evaluated by the Investigator at 7, 15, and 20 minutes post challenge. Mucous discharged was recorded as either absent or present.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: This outcome measure was not assessed for the Vehicle group.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 36 | 36 | 35 | 0
Number analyzed (eyes) | 72 | 71 | 70 | 0
eyes
  7 minutes post-challenge | 7 | 12 | 13 |
  15 minutes post-challenge | 11 | 19 | 18 |
  20 minutes post-challenge | 10 | 16 | 18 |

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | KetoNaph | Ketotifen | Naphazoline | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/35 | 0/37
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/35 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.